CLINICAL TRIAL: NCT05843929
Title: Prevalence of the Appearance of Diabetic Ulcers, After the Manufacture and Adaptation of Personalized Insoles, With Monitoring of Temperature and Plantar Pressure in Diabetic Patients
Brief Title: Prevalence of the Appearance of Diabetic Ulcers in Patients With 3D Insole and LSCI.
Acronym: MYFOOT-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Esther Soler (Other)
Collaborators: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other); Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Sponsor-Investigator, Esther Soler, Principal investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MYFOOT-C-AB/2023
Record Dates: First submitted 2023-03-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diabete Type 2; Diabetic Foot; Neuropathy, Diabetic; Vascular Disease, Peripheral; Diabetic Foot Ulcer
Keywords: Diabete Type 2; Diabetic Foot; Neuropathy, Diabetic; Vascular Disease, Peripheral; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Foot; Diabetic Neuropathies; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients with inclusion criteria and without exclusion criteria will be randomized into two groups with Randomization with sequence concealment, centralized in computer support.
  OxMaR (Oxford Minimization and Randomization) After signing the informed consent, the patients will be divided into two groups.
  1. Group with Laser speckle contrast imaging technique (LSDI), 3D foot creator
  2. Group not LSCI, 3D foot Creator
Masking Description: Open Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group with Laser speckle contrast imaging technique (LSCI) and 3D foot creator use (Experimental): The proposed solution is based on the process synthetized in, and hereafter described:
  * A technician delivers a service at the home of the diabetic patient, who may be subject to different risk of ulcer, with the aim to analyse his/her foot through an integrated set of measurement technologies, based on:
    * the piezoelectric insole that replaces missing pain sensation;
    * Laser speckle contrast imaging technique (LSCI) that measures the blood flow;
    * the multi points temperature device.
  * Data collected by the technician are sent via internet to the reference Hospital or Primary Care Unit where a specialist physician evaluates the acquired information;
  * On the basis of the clinical evaluation and doctor's report on points of foot sensitivity, a 3D model of the foot is created and used by the chiropodist;
  * Using the 3D model of the foot, the chiropodist uses a 3D Editor to design the 3D Model of the insole
  Interventions: Diagnostic Test: LSCI
- Group not use laser speckle contrast imaging technique (LSCI) and not use 3D foot creator use (No Intervention): * The patients of this group will be visited in the hospital:
  * An assessment of the patient's risk of presenting problems due to diabetic foot will be carried out.
  * In this group, the control measures will be established within the usual practice in consultations.
  * No visits will be made to the patient's home. You will always visit the doctor's office.
  * If any problem is detected, the patient will be visited by health personnel and the usual treatments in these patients at present will be applied.

INTERVENTIONS:
Diagnostic Test: LSCI — 1. A technician delivers a service at the home of the patient, who may be subject to different risk of ulcer, with the aim to analyse his/her foot through an integrated set of measurement technologies, based on:a-the piezoelectric insole that replaces missing pain sensation;b- Laser speckle contrast imaging technique (LSCI) that measures the blood flow;c- the multi points temperature device.
  2. Data collected by the technician are sent via internet
  3. On the basis of the clinical evaluation and doctor's report on points of foot sensitivity, a 3D model of the foot is created and used by the chiropodist;
  4. Using the 3D model of the foot, the chiropodist uses a 3D Editor to design the 3D Model of the insole to enable the production of a tailored insole for the patient shoes
  5. The final manufactured insole is then delivered to the patient;
  6. A check survey is periodically carried out by the technician to scan the diabetic foot status progress
  Other Names: 3D FOOT INSOLE
  Arms: Group with Laser speckle contrast imaging technique (LSCI) and 3D foot creator use

SUMMARY:
Diabetes is a serious and chronic disease that affects more than 347 million people in the world. It is the leading cause of death by age and its prevalence is increasing annually throughout the world. Diabetes is a disorder that manifests itself with elevated blood glucose levels that may be the resultof a deficiency in insulin secretion or action, or a combination of both problems.

The "Diabetic foot" includes a number of syndromes in which the interaction of the loss of protective sensation by the presence of sensory neuropathy, the change in pressure points due to motor neuropathy, autonomic dysfunction and decreased Blood flow due to peripheral vascular disease can lead to the appearance of injuries or ulcers induced by minor traumas that go "unnoticed." This situation leads to significant morbidity and a high risk of amputation. It can be prevented with the application of prevention programs, based on the early detection of neuropathy, assessment of associated risk factors, along with the application of a structured program of education and treatment of risk factors.

PRIMARY OBJECTIVES: 1- Comparison of ulceration rates, decrease in amputation rates in the target population with intervention: LSCI, thermography and creation of personalized insoles versus the control group with assessment, treatment and follow-up, without the intervention of interest in the study. 2- Correlation between changes in perfusion and temperature detected in combination of LSCI and thermography to predict diabetic foot ulcers and the risk of having ulcers. Study Model: Parallel Assignment 1:1 . Patients with inclusion criteria and without exclusion criteria will be randomized into two groups with Randomization with sequence concealment, centralized in computer support. OxMaR (Oxford Minimization and Randomization) After signing the informed consent, the patients will be divided into two groups. Number of Arms 2 Masking: None (Open Label) A-GROUP WITH LSCI, 3D FOOT CREATOR FOLLOW UP B- GROUP WITHOUT LSCI, 3D FOOT CREATOR FOLLOW UP.

DETAILED DESCRIPTION:
Regardless of the type of diabetes, failure to achieve optimal glycemic control over time can cause damage to large and small blood vessels, as well as nerves. This damage can affect the function of many body organs and interfere with wound healing. Diabetes is the leading cause of coronary artery disease, and the leading cause of new cases of blindness and kidney disease.

The incidence of foot ulcers in people with diabetes was 2.2% per year, and that having a history of foot ulcers or amputations was strongly associated with the risk of developing foot ulcers in the future.

Prevention of such traumatic events, along with early detection and treatment of foot problems, can reduce the incidence of foot ulceration and amputation. This can be achieved through a risk assessment program, self-care education, and regular reinforcement of that education. Diabetes not only affects the health of individuals but also their families, as well as represents a burden on society.

Research in recent years establishes that reducing contact pressure effectively reduces the incidence of diabetic foot ulcers. In various current scientific studies, methods have been proposed to optimize the distribution of stresses in the contact surfaces between the foot and the template by applying functional gradient structural properties.

Increased skin temperature of the feet is considered to be associated with diabetic peripheral neuropathy, while its decrease is related to the presence of arterial alterations in the foot.

Therefore, there is a higher temperature in the feet of subjects with diabetic peripheral neuropathy, since in diabetic peripheral neuropathy there is an increase in blood flow at the level of the microcirculation. This fact is justified because more heat is dissipated by vasodilation of the arteriovenous shunts, which depend on the control of the sympathetic nerve, causing alterations in thermoregulation. This increase in temperature occurs both on the plantar face and on the dorsal face of the foot, but it is on the back where the temperature increases the most due to the presence of arteriovenous shunts.

When contrasting the data of some publications on this fact, it can be seen how the temperature of the feet of the subjects with Diabetes Mellitus control (without the presence of diabetic peripheral neuropathy) is lower than the temperature of the subjects with Diabetes Mellitus who do present peripheral neuropathy diabetic.

The increase in local temperature is due to the inflammation itself and to the enzymatic autolysis of the tissues, prior to the appearance of an ulceration. An increase in temperature also occurs in subjects with inflammatory processes typical of Charcot arthropathy. The absolute temperatura values of the feet are not considered the best indicators by themselves, since factors such as age, gender or the presence of arteriopathies influence. However, the differences in temperatura between the same point on both feet are relevant, as they are significant at the clinical level.

Specifically, a difference of 2.2º C between the same point on both feet implies a significant/high risk of injury and/or imminent inflammation. The temperature rise may be present for up to a week before an ulcer occurs. If a temperature difference greater than 2.2 ºC is detected but there is no wound/dermal lesion at that point, acute Charcot arthropathy should be considered.

Furthermore, temperature differences correlate with radiological changes and with markers of bone remodeling. The rise in temperature is usually too subtle to be detected manually, so it is measured.

Currently, three temperature measurement systems are used, which are applied through two types of techniques: thermography and thermometry. Thermography tests are classified into infrared and thermosensitive liquid crystal overlays. Thermometry tests are divided into infrared and termal sensors.

Why assess the temperature of the feet in Diabetes Mellitus? Diabetic ulcers generate a high economic cost, a high personal burden and carry an important social significance, both the process in which the injury is present and after the amputation suffered after a disastrous evolution of it.

However, its prevention is simple, economical and based on scientific evidence that supports it.

Prevention has a great impact since 75% of plantar ulcers can be prevented. Despite this, for every euro spent on prevention of plantar ulcers due to Diabetes Mellitus, 10 euros are used to cure them. One thing to keep in mind is that after the appearance of the first plantar ulcer in a patient with Diabetes Mellitus, the risk of recurrence is between 30-87% due to NPD. The arguments that justify the inclusion of thermal assessment in the neurological examination protocols of the feet of subjects with Diabetes Mellitus are the following: 1. First of all, the investigators must consider that the prevention of Diabetic Foot, it is currently based on exploration using two qualitative sensory tests with the Semmens-Weinstein 5.07 monofilament and the Rydel-Scheiffer 128 Hz graduated tuning fork, self-inspection by the patient and pulse palpation, not being the exploration of the temperature included. Effectiveness of preventive interventions for the appearance of ulcers in Diabetes Mellitus, being more effective the measurement of the temperature of the skin of the feet (once a day), advice and preventive footwear. These authors reinforce the suggestion of including temperatura measurement due to the short time of application in the exploratory screening with respect to preventive footwear. The importance of the heat resistance of the sole materials of footwear in subjects with Diabetes Mellitus is relevant since thermal perception is altered in them, and it must be taken into account that a temperature greater than 44º C generates a burn in the skin, with a temperature of 55º C, the burn occurs in 20 seconds and while, if the temperature is greater tan 60º C, only 3 seconds are needed for the burn to develop. Self-monitoring of temperatura (assessment of the same point in 2 feet) decreases the rate of appearance of ulcers.

There is a temperature interval, a difference of 2.2ºC between the two feet, which is used to control the appearance of lesions typical of Diabetic Foot. This interval, as a diagnostic test for infection, has a specificity of 25% and a sensitivity of 80% 40. With a temperature difference range of 1.35ºC, it is considered that urgent action is necessary28. Another argument is that the evaluation of the temperature of the feet is an effective and non-invasive technique. Its applicability is viable. Thermography is useful in detecting plantar ulcers with osteomyelitis. At a practical level, temperature control is an effective parameter to control bone consolidation and the evolutionary process of Charcot's disease, allowing a safe removal of immobilization.

The tendency to evaluate this parameter may be instruments with automatic storage of the processed data, with immediate obtaining of the calculation of the temperature differences The conclusions of this work are the following:

1. A difference of 2.2ºC at the same point on both feet of a subject indicates the appearance of lesions typical of Diabetic Foot, either ulceration if there is a lesion, or Charcot arthropathy.
2. The measurement of the temperature of the feet can be done by thermography and thermometry.
3. Scientific evidence indicates that controlling the temperature of the feet decreases the rate of ulcerations in Diabetes Mellitus.
4. The investigators advocate the inclusion of thermal assessment in the exploration protocol of subjects with Diabetes Mellitus, due to its effectiveness in preventing ulcerations as well as its short screening time.

Level of evidence related to the mechanism of action of the intervention in the planned clinical study population Diabetic foot ulcers (DFU) are a frequent complication, produced by sensory neuropathy and mechanical stress, it has been shown that the maximum plantar pressure (PPM) and the máximum pressure gradient (PPG) during walking are determining factors of these ulcers. In the clinical trial by Fernando ME et al., conducted in Australia, they evaluated plantar pressures in patients with active DFUs compared with patients with diabetes without a history of DFUs (diabetes controls) and people without diabetes (healthy controls), compared to those with 16 cases and 63 controls underwent plantar pressure measurement using an in-shoe pressure measurement software called Footscan® (F-scan), the cases had higher PPM in several sites: in the hallux, metatarsals and region midfoot compared to controls at follow-up. Plantar pressures assessed during walking were higher in patients with diabetes with UPD chronic than controls at various plantar sites, therefore offloading (relieving pressure) is necessary in patients with DFUs to facilitate healing.

ELIGIBILITY:
Inclusion Criteria:

1. The sample will include all the people who sign the informed consent.
2. Patients aged between 18 and 80 years.
3. Patients diagnosed with Diabetes Mellitus (more than 5 years from diagnosis), from the Department of Health Elche Hospital General.
4. Patients with Risk Level 2 and 3 according to the International Working Group on the Diabetic Foot - IWGDF.

Exclusion Criteria:

1. People who do not give their consent to participate in the study.
2. Patients who have previously had treatment with plantar orthoses or personalice insole.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The ankle-brachial index (ABI) | 15 minutes
  The ankle-brachial index (ABI). The test compares the blood pressure in the ankle and the blood pressure in the arm. The provider uses a blood pressure cuff and an ultrasound device.
  The normal result of the ABI is 1.00 or more. If you have an ABI of less than 0.90 at rest, you probably have PAD. An ABI of less than 0.40 is a sign of severe PAD. If there are problems with the arteries in your ankle, your provider may measure your toe-brachial index (BPI), which measures blood pressure in your big toe. A BDI of less than 0.7 is abnormal.
Laser speckle contrast imaging technique (LSCI) that measures the blood flow | 15 minutes
  the Laser Speckle Contrast Imaging (LSCI) technology, also known as the Laser Speckle Imaging system (LSI), which is non-invasive with non-contact, high time resolution, high spatial resolution, and full-field rapid imaging. It provides real-time dynamic blood flow monitoring and recording methods for research in life sciences
Design the 3D model of the insole | 2 day
  Custom 3D-printed orthotic insoles. Translate foot measurement data into 3D-printed orthotics that fit the individual's foot perfectly.
Diabetic foot exam:neurologic examination-PAINFUL AND TACTILE SENSITIVITY | 15 minutes
  * The patient will be placed in supine position.
  * The tests will be performed alternating the exploration of painful and tactile sensitivity until completing all the sections.
  Execution:
  * Instruct the patient to close their eyes.
  * Alternate touches with the pointed object and cotton on the planting areas (A-F) and on the dorsal areas (G-I) indicated in the drawings.
  * You have to wait a minimum of 2 seconds between touches to avoid the summation effect.
  * Do not perform the scan in areas with hyperkeratosis or calluses.
  Interpretation
  - Yes (Painful): , when the patient communicates to the clinician the sensation of puncture in the explored area.
Diabetic foot exam:neurologic examination-VIBRATORY SENSITIVITY | 15 minutes
  * The patient will be placed in supine position.
  * The tests will be performed alternating the exploration of painful and tactile sensitivity until completing all the sections.
  * Instruct the patient to close their eyes.
  * Alternate touches with the pointed object and cotton on the planting areas (A-F) and on the dorsal areas (G-I) indicated in the drawings.
  * You have to wait a minimum of 2 seconds between touches to avoid the summation effect.
  * Do not perform the scan in areas with hyperkeratosis or calluses. Interpretation
  * No (Painful): When the patient does not communicate to the clinician the sensation of puncture in the explored area.
  * No (Tactyl): When the patient does not communicate to the clinician the sensation of contact in the explored area.
Diabetic foot exam:neurologic examination-THERMAL SENSITIVITY | 15 minutes
  1. Previous Considerations:
     * This test may be skipped if the pain sensitivity is normal.
     * Previously, both stimuli must be performed in another uncommitted area of the body.
     * 2 test tubes will be prepared with water at two different temperatures: 1 tube called 'cold' with the water at a temperature below 15ºC and 1 tube called 'hot' with the water at a temperature above 40ºC.
  2. Execution:
     * Instruct the patient to close their eyes.
     * The 'hot' and 'cold' tube will be applied to the skin of the dorsal area (G-I) randomly.
     * Ask the patient if the sensation perceived after the application of a tube (cold or hot), is of higher or lower temperature than the tube previously applied.
     * Randomly toggle between the G-I zones marked on the chart.
  3. Interpretation:
     * Cold: When the patient communicates to the clinician the feeling of cold.
     * Hot: When the patient does not communicate to the clinician the sensation of heat.
Diabetic foot exam:neurologic examination-PROTECTIVE SENSITIVITY | 15 minutes
  1. Execution:
     * Instruct the patient to close their eyes.
     * Apply the monofilament randomly on the A-F zones of the sole of the foot and at the points of the dorsal zone G-I, pressing until the filament bends.
     * Hyperkeratostic areas should be avoided.
  2. Interpretation:
     * Yes: When the patient communicates to the clinician the sensation of the stimulus.
     * No: When the patient does not communicate to the clinician the sensation of the stimulus.
Diabetic foot exam:neurologic examination- ARTHROKINETIC SENSITIVITY | 15 minutes
  1. Execution:
     * The test must be performed previously on a finger of the hand, so that the patient understands the performance of the test.
     * The patient will close the eyes and move the distal phalanges of the 1st, 3rd and 5th toes, a few degrees towards dosal flexion and plantar flexion.
     * The patient will be asked in which direction the joint has moved.
  2. Interpretation:
     * Yes: When the patient correctly communicates the direction of movement.
     * No: When the patient does not communicate correctly the direction of movement.
Diabetic foot exam: musculoskeletal examination | 10 minutes
  A method of evaluating muscle strength is the Medical Research Council Manual Muscle Testing Scale.This method involves testing key muscles from the upper and lower extremities against gravity and the examiner's resistance and grading the patient's strength on a 0 to 5 scale.
  * Hallux Valgus: The test will be performed by visualization. Interpretation: It will be evaluated following the criteria of the Manchester Scale for the graduation of the Hallux Abductus Valgus (Garrow AP, Papageorgiou A, Silman AJ, Thomas E, Jayson MI, Macfarlane GJ. The grading of hallux valgus. The Manchester Scale. J Am Podiatr Med Assoc. 2001;91(2):74-78. doi:10.7547/87507315-91-2-74) in; A: Normal. B: Mild. C: Moderate. D: Severe
  * Hallux Extensus.
  * Hallux Flexus. https://wtcs.pressbooks.pub/nursingskills/chapter/13-4-musculoskeletal-assessment/
Diabetic foot exam: dermatologic examination | 10 minutes
  All the test will be performed by visualization. - Hyperkeratosis.-Ulcer shall be considered to be the total loss of the epidermis.-Onychocryptosis shall be considered to be the incrustation of the lateral edges of the nail.-Onychogriphosis shall be considered to be the thickening of the nail plate with a hyperkeratotic.-Onychomycosis is considered to be any nail infection caused by any fungus. -Hyperhidrosis will be considered the excessive increase in sweating of the feet.-Anhidrosis will be considered to be the absence or decrease of sweating of the feet.-Signs of infection will be considered to be the presence of red, hot, sensitive and indurated skin with the presence of pain in the area. Dermatomycosis.-A circumscribed dermatological lesion greater than 1 cm and with liquid content.-Hematoma will be considered to be a hemorrhage circumscribed in the skin.-A linear disruption of the stratum corneum shall be considered a fissure.

SECONDARY OUTCOMES:
Diabetes Self-Care | 10 minutes
  A psychometric analysis of the Self-Care Inventory-revised with adults. TEST: Self-Care Inventory-revised (SCI-R) The SCI-R is a brief, psychometrically sound measure of perceptions of adherence to recommended diabetes self-care behaviors of adults with type 1 or type 2 diabetes.
  Weinger, K., Butler, H. A., Welch, G. W., & La Greca, A. M. (2005). Measuring diabetes self-care: a psychometric analysis of the Self-Care Inventory-Revised with adults. Diabetes care, 28(6), 1346-1352. https://doi.org/10.2337/diacare.28.6.1346

CONTACTS AND LOCATIONS:
Overall Officials: ESTHER SOLER, BSN, Principal Investigator — CGE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sibbald RG, Mufti A, Armstrong DG. Infrared skin thermometry: an underutilized cost-effective tool for routine wound care practice and patient high-risk diabetic foot self-monitoring. Adv Skin Wound Care. 2015 Jan;28(1):37-44; quiz 45-6. doi: 10.1097/01.ASW.0000458991.58947.6b. PMID 25502975
- [Background] Pallin JA, Van Netten JJ, Kearney PM, Dinneen SF, Buckley CM. Do we screen, examine or assess to identify the "at-risk" foot in diabetes-time for agreed terms and definitions? Diabet Med. 2023 Jan;40(1):e14976. doi: 10.1111/dme.14976. Epub 2022 Oct 26. No abstract available. PMID 36251428
- [Background] Garcia-Madrid M, Garcia-Alvarez Y, Sanz-Corbalan I, Alvaro-Afonso FJ, Lopez-Moral M, Lazaro-Martinez JL. Predictive value of forefoot plantar pressure to predict reulceration in patients at high risk. Diabetes Res Clin Pract. 2022 Jul;189:109976. doi: 10.1016/j.diabres.2022.109976. Epub 2022 Jun 27. PMID 35772587
- [Result] Ahmed H, Elshaikh T, Abdullah M. Early Diabetic Nephropathy and Retinopathy in Patients with Type 1 Diabetes Mellitus Attending Sudan Childhood Diabetes Centre. J Diabetes Res. 2020 Nov 24;2020:7181383. doi: 10.1155/2020/7181383. eCollection 2020. PMID 33299891
- [Result] Norhammar A, Malmberg K, Diderholm E, Lagerqvist B, Lindahl B, Ryden L, Wallentin L. Diabetes mellitus: the major risk factor in unstable coronary artery disease even after consideration of the extent of coronary artery disease and benefits of revascularization. J Am Coll Cardiol. 2004 Feb 18;43(4):585-91. doi: 10.1016/j.jacc.2003.08.050. PMID 14975468
- [Result] Valk GD, Kriegsman DM, Assendelft WJ. Patient education for preventing diabetic foot ulceration. A systematic review. Endocrinol Metab Clin North Am. 2002 Sep;31(3):633-58. doi: 10.1016/s0889-8529(02)00021-x. PMID 12227125
- [Result] Bus SA, Armstrong DG, Gooday C, Jarl G, Caravaggi C, Viswanathan V, Lazzarini PA; International Working Group on the Diabetic Foot (IWGDF). Guidelines on offloading foot ulcers in persons with diabetes (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3274. doi: 10.1002/dmrr.3274. PMID 32176441
- [Result] Bus SA. Innovations in plantar pressure and foot temperature measurements in diabetes. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:221-6. doi: 10.1002/dmrr.2760. PMID 26467347
- [Result] Liu C, van Netten JJ, van Baal JG, Bus SA, van der Heijden F. Automatic detection of diabetic foot complications with infrared thermography by asymmetric analysis. J Biomed Opt. 2015 Feb;20(2):26003. doi: 10.1117/1.JBO.20.2.026003. PMID 25671671
- [Result] van Netten JJ, Price PE, Lavery LA, Monteiro-Soares M, Rasmussen A, Jubiz Y, Bus SA; International Working Group on the Diabetic Foot. Prevention of foot ulcers in the at-risk patient with diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:84-98. doi: 10.1002/dmrr.2701. PMID 26340966
- [Result] Clifton T, Khoo TW, Andrawos A, Thomson S, Greenwood JE. Variation of surface temperatures of different ground materials on hot days: Burn risk for the neuropathic foot. Burns. 2016 Mar;42(2):453-6. doi: 10.1016/j.burns.2015.08.026. Epub 2016 Jan 12. PMID 26797153
- [Result] Lung CW, Wu FL, Liao F, Pu F, Fan Y, Jan YK. Emerging technologies for the prevention and management of diabetic foot ulcers. J Tissue Viability. 2020 May;29(2):61-68. doi: 10.1016/j.jtv.2020.03.003. Epub 2020 Mar 17. PMID 32197948
- [Result] Fernando ME, Crowther RG, Lazzarini PA, Yogakanthi S, Sangla KS, Buttner P, Jones R, Golledge J. Plantar pressures are elevated in people with longstanding diabetes-related foot ulcers during follow-up. PLoS One. 2017 Aug 31;12(8):e0181916. doi: 10.1371/journal.pone.0181916. eCollection 2017. PMID 28859075
- [Result] Yang L, Wu Y, Zhou C, Xie C, Jiang Y, Wang R, Ye X. Diabetic foot ulcer risk assessment and prevention in patients with diabetes: a best practice implementation project. JBI Evid Implement. 2022 Dec 1;20(4):269-279. doi: 10.1097/XEB.0000000000000306. PMID 35013076
- See also: EUROPA INFORMED CONSENT INFORMATION — https://ec.europa.eu/research/participants/data/ref/fp7/89807/informed-consent_en.pdf
- See also: IWGDF GUIDELINES — https://iwgdfguidelines.org/about-iwgdf-guidelines/iwgdf-now/